CLINICAL TRIAL: NCT00162331
Title: AIR-MI: Assessment of Ischemia and Remodeling Following Acute Myocardial Infarction
Brief Title: CARDIOLITE-413: A Study for Patients Who Had a PCI for an Acute MI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Qi Zhu, MD Sr. Medical Director, Lantheus Medical Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARDIOLITE-413
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Technetium Tc99m Sestamibi

SUMMARY:
The purpose of this clinical study is to learn if there are any changes in how blood gets to your heart muscle and if your heart size changed after your heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary or rescue PCI for acute MI with ECG evidence of a large territory at risk.

Exclusion Criteria:

* History of prior MI or CABG surgery, persistent LBBB, Atrial Fibrillation, End stage renal disease, Weight > 350 lbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To better understand the interactions between the abnormalities in blood supply from the small vessels of the heart to the heart muscle after a heart attack and the changes in heart size 6 months after the heart attack.

SECONDARY OUTCOMES:
To estimate the frequency of residual ischemia as assessed by stress myocardial perfusion imaging (MPI) in patients undergoing primary PCI for AMI.
To estimate the 6-month cardiac event rates (composite of death, another heart attack, hospitalization for heart failure, and irregular heart beats requiring treatment).
To determine the relationship between changes (from baseline) in LV systolic volume index and LVEF, as measured by gated SPECT imaging 6 months following reperfusion, and the presence and severity of residual ischemia.
To measure the performance of angiographic parameters of success of reperfusion therapy (TIMI frame count and TIMI myocardial perfusion grade) in predicting the presence of residual ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhu, MD, Study Director — Lantheus Medical Imaging
Locations (8):
- United States (4):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Boston, Massachusetts
  - Local Institution, Nashville, Tennessee
  - Local Institution, Seattle, Washington
- Brazil (2):
  - Local Institution, Curibita
  - Local Institution, São Paulo
- Canada (2):
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario